CLINICAL TRIAL: NCT06874439
Title: An Evaluation of the WHO QUAlityRights Program
Acronym: EQUAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS-CCOMS (Other)
Collaborators: INSERM ECEVE 1123 (Unknown); L'Assistance Publique - Hopitaux de Paris (AP-HP) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-A00092-45; PREPS-22-0042 (Other Grant/Funding Number: French Ministry of Health)
Record Dates: First submitted 2025-02-20; First posted 2025-03-13 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Recovery; Organization of Health Service; Mental Health Care; Mental Health Services
Keywords: User rights; Recovery-oriented practices; Mental Health Settings; Satisfaction with care; Interventional study; Randomized controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Sectors receiving the WHO QualityRights program
  Interventions: Other: WHO QualityRights program
- Usual practices (No Intervention): Sectors not receiving the WHO QualityRights program, and maintaining usual practices

INTERVENTIONS:
Other: WHO QualityRights program — The WHO's QualityRights program involves an assessment, called observation, of mental health care services by an ephemeral multidisciplinary team, which provides feedback and recommendations for improving care practices. The observation team, trained in the QualityRights (QR) methodology, includes mental health professionals, researchers, legal experts, and management staff from mental health organizations. Each team always incorporates at least one expert by experience and one informal caregiver or family member. Participation in the program is voluntary and initiated at the request of healthcare facilities.
  The observation is structured into three stages:
  1. Site preparation
  2. On-site observation
  3. Restitution of observation report and follow-up
  Arms: Intervention

SUMMARY:
The World Health Organization's (WHO) QualityRights (QR) program offers assessments and recommendations to help mental health facilities, on a voluntary basis, improve their care practices towards better respect of the rights of service users. The aim of this study is to evaluate the QR program in a French national context.

The main questions it aims to answer are:

* Does the QR program improve perceived satisfaction with care among mental health service users?
* What are the implementation procedures of the program?
* What is its budgetary impact?

Researchers will compare the QR program intervention with usual practices.

DETAILED DESCRIPTION:
In France, despite the existence of recommendations and a restrictive legal framework, the use of restraint practices in psychiatry remains widespread, and the duration and conditions of hospitalization do not always guarantee respect for users' rights.

The World Health Organization's (WHO) QualityRights (QR) program offers assessments, called "observations", and recommendations to help mental health facilities, on a voluntary basis, improve their care practices towards better respect of the rights of service users. However, the program has never been evaluated in a French national context.

The WHO QR program, published in 2012 and regularly updated since, aims to improve the quality of care in mental health and related services and promote the rights of people with psychosocial, intellectual and cognitive disabilities.

The reference base for the tools that make up the program is the United Nations Convention on the Rights of Persons with Disabilities (CRPD), ratified by France in 2010. This international convention defines ambitious objectives in terms of respect for rights, some of which are particularly relevant to mental health services. However, the convention does not offer any concrete indications as to how these major international standards are to be applied.

The QR program provides a concrete response to this need, offering observation and training tools not only for mental health services, but more broadly for all those concerned by mental health issues. In particular, the observation methodology is designed to respond to a request for support in changing practices that comes directly from a facility.

The WHO Collaborating Centre in Lille is mandated by the WHO to roll out this program in France and other French-speaking countries. It is expected that the QualityRights approach will act as a lever for change in the organization of services, providing a multidisciplinary perspective on users' rights and recovery-oriented practices.

The primary research objective is to evaluate the effectiveness of the QR program on the perceived satisfaction with care of mental health service users.

The secondary research objectives concern:

A. Evaluating the effectiveness of the QR program on:

1. Improving work-related quality of life among mental health professionals
2. Decreasing the number of involuntary admissions
3. Reducing the length of full-time hospital stays
4. Reducing the number of acts of seclusion and restraint
5. The distribution of clinical activity in favour of ambulatory activity

B. Evaluating the efficiency and the budgetary impact of the QR program.

C. Conducting an implementation study to understand the appropriation of the recommendations by professionals and management following the introduction of the QR program by exploring the representations linked to the QR program and respect for users' rights among mental health professionals.

This research involves an effectiveness study, supplemented by an implementation study based on a qualitative methodology, and an economic evaluation.

The effectiveness study is a cluster randomized trial designed to compare the effectiveness of the QR program intervention versus usual practices on user satisfaction. The cluster is defined at the level of the psychiatric sector (the public psychiatric care entity organizing the mental health care of a population within a pre-specified geographical and demographic area in France, to meet local needs). 10 psychiatric sectors are participating, randomized into two groups: the intervention group receiving the QR program and the control group maintaining their usual practices.

Data will be collected in both groups at baseline, and during follow-up at 1 and 2 years. The implementation study and the economic evaluation will be carried out in the intervention group after the effectiveness study.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* Persons having formulated a non-opposition to participate in the study
* Population a (users): Service users of the psychiatric sectors involved in the study hospitalized full-time since at least 3 days in an inpatient unit.
* Population b (professionals): Mental health professionals working in the sector since at least 3 months at the time of study participation

Exclusion Criteria:

* Persons physically or psychologically unable to participate at the time of the study
* Persons subject to a safeguard of justice measure
* Persons who do not speak or understand the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with care | At baseline, at 1 year, and at 2 years
  Service user satisfaction with care score assessed using the Verona Service Satisfaction Scale (VSSS-54F)

SECONDARY OUTCOMES:
Work-related quality of life | At baseline, at 1 year, and at 2 years
  Work-related quality of life score for mental health professionals assessed using the SERENAT scale
Involuntary psychiatric hospitalisations | At baseline, at 1 year, and at 2 years
  Number of involuntary hospitalizations in the 6 months preceding the time point
Length of stay | At baseline, at 1 year, and at 2 years
  Length of stay for each patient in the 6 months preceding the time points
Seclusion and restraint | At baseline, at 1 year, and at 2 years
  Number of acts of seclusion and restraint in the 6 months preceding the time points
Distribution of hospital activity | At baseline, at 1 year, and at 2 years
  Hospital case load and outpatient service utilization in the 6 months preceding the time points
Cost-utility | 24 months
  Incremental cost-utility ratio in cost per QALY gained (EQ-5D-5L questionnaire)
Cost-effectiveness | 24 months
  Incremental cost-effectiveness ratio in cost per VSSS-54F score points gained
Budgetary impact - costs | 5 years after hypothetical generalization
  Costs associated with the generalization of the QR program
Budgetary impact - QALY | 5 years after hypothetical generalization
  The number of QALYs will be calculated with and without the QR program to assess the gains associated with its generalization.
Budgetary impact - Involuntary psychiatric hospitalizations | 5 years after hypothetical generalization
  The number of involuntary hospitalizations will be calculated with and without the QR program to assess the gains associated with its generalization.
Budgetary impact - Length of stay | 5 years after hypothetical generalization
  The length of stay will be calculated with and without the QR program to assess the gains associated with its generalization.
Budgetary impact - Seclusion and restraint | 5 years after hypothetical generalization
  The number of acts of seclusion and restraint will be calculated with and without the QR program to assess the gains associated with its generalization.
Implementation | In the 1 year following the last time point
  Qualitative methods will be used through semi-structured interviews conducted with 10 mental health professionals per sector of the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Déborah Sebbane, MD, PhD, Study Chair — GCS-CCOMS & ECEVE 1123 INSERM
Locations (10):
- France (10):
  - Public mental health establishment of Lille Metropole (59G09/G10), Armentières
  - Public mental health establishment of Lille Metropole (59G20), Armentières
  - Hospital Centre of Erstein, Erstein
  - Psychotherapeutic Center of Nancy, Laxou
  - Hospital Centre Drôme Vivarais, Montéléger
  - Hospital Care Center of Nanterre, Nanterre
  - Hospital Centre Sainte-Marie Nice, Nice
  - Hospital Center of Plaisir (78G16), Plaisir
  - Hospital Center of Plaisir (78G18), Plaisir
  - Hospital Center of Candélie, Pont-du-Casse

IPD SHARING:
Plan to Share IPD: No